CLINICAL TRIAL: NCT00146926
Title: Comparison of Three Different Strategies to Prevent Propofol Induced Pain During Infusion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2004.367
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Induction of Total Intravenous General Anesthesia
Keywords: Propofol; pain; general anesthesia; prevention
MeSH Terms: conditions — Pain | interventions — Ketamine; Ephedrine; Lidocaine

INTERVENTIONS:
Drug: kétamine 20mg
Drug: ephedrine 3mg
Drug: lidocaine 40mg

SUMMARY:
Propofol is a popular intravenous drug to induce anesthesia but it causes local pain with an incidence between 40 and 90%. Three different strategies to prevent propofol induced pain will be studied compared with placebo. Pain will be scored with a four-point scale.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults (ASA 1-2) for scheduled surgery under general anesthesia with propofol

Exclusion Criteria:

* pregnant
* sedative or analgesic drug 24h before surgery
* allergy with drug used in the study
* difficulty of communication
* absence of informed written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-09

PRIMARY OUTCOMES:
After prophylactic solution, evaluation of the pain caused by injection of propofol with a four-point scale before lose of consciousness

SECONDARY OUTCOMES:
Explicite and implicite memory of pain immediately after surgery and on day one
Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Vincent PIRIOU, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Grégoire CHATAIN, Lyon, France